CLINICAL TRIAL: NCT02948114
Title: The Effect of Feeding Infant Formula Containing Prebiotics and/or Probiotics
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment challenges
Sponsor: Mead Johnson Nutrition (Industry)
Collaborators: Beijing Kangchen Technologies (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 6026
Record Dates: First submitted 2016-10-26; First posted 2016-10-28 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Metabolomics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Control: Cow milk-based infant formula (Active Comparator): Cow milk-based infant formula
  Interventions: Other: Control: Cow milk-based infant formula
- Experimental 1: Cow milk-based infant formula (Experimental): Cow milk-based infant formula with prebiotics
  Interventions: Other: Experimental 1: Cow milk-based infant formula
- Experimental 2: Cow milk-based infant formula (Experimental): Cow milk-based infant formula with probiotics
  Interventions: Other: Experimental 2: Cow milk-based infant formula
- Experimental 3: Cow milk-based infant formula (Experimental): Cow milk-based infant formula with prebiotics and probiotics
  Interventions: Other: Experimental 3: Cow milk-based infant formula
- Human Milk Reference (No Intervention): Human Milk Reference

INTERVENTIONS:
Other: Control: Cow milk-based infant formula
  Arms: Control: Cow milk-based infant formula
Other: Experimental 1: Cow milk-based infant formula — Experimental 1: Cow milk-based infant formula with prebiotics
  Arms: Experimental 1: Cow milk-based infant formula
Other: Experimental 2: Cow milk-based infant formula — Experimental 2: Cow milk-based infant formula with probiotics
  Arms: Experimental 2: Cow milk-based infant formula
Other: Experimental 3: Cow milk-based infant formula — Experimental 3: Cow milk-based infant formula with prebiotics and probiotics
  Arms: Experimental 3: Cow milk-based infant formula

SUMMARY:
The study is intended to evaluate the microorganisms found in infant stools when consuming study formulas containing prebiotics and/or probiotics compared to infants consuming mother's own breast milk.

ELIGIBILITY:
Inclusion Criteria:

* Singleton, 10-14 days of age at registration/randomization
* Term infant with birth weight of 2500 grams or more from a vaginal birth
* Formula feeding infants must be on formula for at least 3 days
* Human milk fed infants must have received mother's own breast milk from 1 day of age to study registration and mother has intention to exclusively provide mother's own breast milk for the duration of the study
* Signed informed consent

Exclusion Criteria:

* History of underlying metabolic or chronic disease or immune compromised
* Feeding difficulties or formula intolerance

Ages: 10 Days to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change in fecal microbiota | 3.5 months

SECONDARY OUTCOMES:
Body Weight measured at each study visit | Up to 3.5 months
Body Length measured at each study visit | Up to 3.5 months
Head circumference measured at each study visit | Up to 3.5 months
Recall of infant formula usage at each study visit | Up to 3.5 months
Recall of gastrointestinal tolerance questionnaire at each study visit | Up to 3.5 months
Medically-confirmed adverse events collected throughout the study period | Up to 3.5 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven Wu, Study Director — Mead Johnson Nutrition
Locations (1):
- Hainan Province Women & Children Hospital, Haikou, Hainan, China